CLINICAL TRIAL: NCT01837693
Title: HPV as Primary Screening Test in Cervical Cancer Prevention: From DNA to mRNA? A Randomised Controlled Trial Nested in a Double Testing Study With Long Term Follow up
Brief Title: Cervical Cancer Prevention: From DNA to mRNA? - New Technologies for Cervical Cancer Screening 2
Acronym: NTCC2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda USL Reggio Emilia - IRCCS (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: cervicalscreening_mRNA_p16
Record Dates: First submitted 2013-04-18; First posted 2013-04-23 (Estimated); Last update posted 2025-06-26 (Actual); Status verified 2017-06

CONDITIONS: Precancerous Conditions; Neoplasms
Keywords: cervical cancer screening; CIN; cervical cancer; biomarkers; sensitivity and specificity
MeSH Terms: conditions — Precancerous Conditions; Neoplasms; Uterine Cervical Neoplasms; Hypersensitivity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | US Export: No

ARMS (2):
- one year follow up (No Intervention): A random sample of HPV positive women with negative cytology will be invited to repeat HPV DNA test and biomarkers after a year, as recommended by the current screening protocols based on HPV DNA
- direct sending in colposcopy (Experimental): Experimental: immediate colposcopy. A random sample of HPV positive women with negative cytology will be sent to immediate colposcopy
  Interventions: Procedure: Experimental: immediate colposcopy

INTERVENTIONS:
Procedure: Experimental: immediate colposcopy — A immediate colposcopy in this arm may detect potentially spontaneous regressive cervical lesions, so may determine an over diagnosis and over treatment, which the study want to estimate
  Arms: direct sending in colposcopy

SUMMARY:
In industrialized countries, cervical cancer is a well controlled disease thanks to the diffusion of Pap test and, in particular, to organized screening programs, which are able to detect and treat pre-invasive lesions (cervical intraepithelial neoplasia, CIN). The human papilloma virus (HPV) has been recognised as the necessary, but not sufficient, cause of cervical cancer, so a new screening test based on the identification of high risk (HR) HPV types has been developed(HPV DNA test). This test has demonstrated to be more effective than cytology in reducing the incidence and the mortality of cervical cancer, but it is less specific, so the use of a test triage is necessary to reduce the number of colposcopies and the risk of over-diagnosis (due to the potential regressivity of pre-invasive lesions). Until now, the triage test used is the cytology (Pap test).

Recently specific biomarkers (mRNA and p16 tests) have been introduced for high grade CIN, targeting the molecular alterations strictly associated to transformation rather than simply detecting HR-HPV infections. These tests are more specific than HPV DNA test with a modest reduction of sensitivity for high-grade lesions.

This is a multicenter randomised trial nested into some Italian screening programs based on the use of HPV DNA test as primary test.

All women with positive HPV DNA test will be tested for cytology and also for mRNA and p16. Women with positive cytology will be referred to colposcopy, while women with negative cytology will be randomized into two arms.

This study aims to evaluate if mRNA and p16 could be used as test of triage of HPV DNA or as a primary screening test with direct sending in colposcopy.

In particular the main objectives are:

* Measuring the cumulative detection rate of CIN2+ in the five years following a HPV DNA positive test and mRNA or p16 negative.
* Measuring the potential reduction of overdiagnosis of using mRNA or p16 test instead of DNA, with direct sending in colposcopy
* Measuring the reduction of overdiagnosis of cytological triage or triage with mRNA or p16 compared to the direct sending in colposcopy in women with HPV DNA test positive.

Secondary objectives are:

* to assess the feasibility of mRNA testing in primary screening
* to validate the sample techniques for the new tests
* to standardize quality controls for the the new tests

DETAILED DESCRIPTION:
Individual data about the following study steps are collected according a fixed format:

1. recruited women
2. HPV DNA result
3. cytology and randomization results
4. p16 result
5. mRNA result
6. colposcopies (with relative cytology and histologies) results
7. Women excluded after informed consent
8. Interventions During the first year of recruitment, there will be two semi-annual sending of data, then each year.

To analyze the study progress in each center, summary tables will periodically send to the PI.

All CIN lesions and cancers found in the study will be be blindly reviewed. A set of quality assurance procedures will be implemented for both the molecular tests, including the use of controls provided by the manufacturers with known HPV DNA or mRNA content and the circulation of clinical samples prepared by the laboratories participating in the study.

ELIGIBILITY:
Inclusion Criteria:

* women invited for a new screening round based on HPV DNA test

Exclusion Criteria:

* women not resident in the screening area, or pregnant, or with treated CIN in the 5 previous years, or in post-colposcopy follow up, or in repetition for unsatisfactory cytology.

Ages: 25 Years to 59 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 41127 (Actual)
Dates: Start 2013-06-01 (Actual); Primary Completion 2017-01-01 (Actual); Study Completion 2017-01-01 (Actual)

PRIMARY OUTCOMES:
cumulative incidence of CIN2+ in women with positive DNA and negative mRNA or p16 | 5 years
  Sum of CIN2+ detected in women with positive DNA and negative mRNA or p16 tests during the entire period (5 years) divided by the total number of CIN2+ found in the study. The HPV DNA test will be the final follow-up test, since it is the most sensitive test among the candidates for screening, so it is the one that allows to estimate more accurately the prevalence of lesions.

SECONDARY OUTCOMES:
comparison between CIN2+ detection rates in the two arms in women with p16 or mRNA negative | 1 year
  proportion of CIN2+, HPV DNA positive and p16 or mRNA negative, which regress in a year
comparison between CIN2+ detection rates in the two arms in women with negative cytology | 1 year
  measure of how much the cytological triage can reduce overdiagnosis compared to HPV DNA with direct sending to colposcopy
comparison between CIN2+ detection rate in the two arms in women with p16 or mRNA positive | 1 year
  direct comparison of the effectiveness between a screening based on the HPV mRNA or p16 test followed by cytological triage and a screening with direct sending to colposcopy

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Giorgi Rossi, PhD, Principal Investigator — Epidemiology Service, Local Health Authority of Reggio Emilia, Italy
Locations (5):
- Italy (5):
  - Unità Locale Socio-Sanitaria 17 Este Monselice, Este
  - Istituto per lo Studio e la Prevenzione Oncologica, Florence
  - Azienda Sanitaria Locale 2- Regione Umbria, Perugia
  - Azienda Sanitaria della Provincia Autonoma di Trento, Trento
  - Centro per la Prevenzione Oncologica del Piemonte, Turin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Del Mistro A, Mancuso P, Carozzi F, De Marco L, Bisanzi S, Pompeo G, Ronco G, Gori S, Allia E, Gustinucci D, Frayle H, Iossa A, Cesarini E, Bulletti S, Passamonti B, Viti J, Toniolo L, Venturelli F, Giorgi Rossi P, Benevolo M; NTCC2 Working Group. Impact of differentiating between persistent and new infections on colposcopy referral in HPV-positive triage-negative women: results from the NTCC2 study. Infect Agent Cancer. 2025 Nov 20;20(1):84. doi: 10.1186/s13027-025-00713-8. PMID 41261407
- [Derived] De Marco L, Bisanzi S, Ronco G, Mancuso P, Carozzi F, Allia E, Rizzolo R, Gustinucci D, Frayle H, Viti J, Iossa A, Cesarini E, Bulletti S, Passamonti B, Gori S, Toniolo L, Venturelli F, Del Mistro A, Giorgi Rossi P, Benevolo M; NTCC2 Working Group. Extended HPV genotyping by the BD Onclarity assay: concordance with screening HPV-DNA assays, triage biomarkers, and histopathology in women from the NTCC2 study. Microbiol Spectr. 2025 Jan 7;13(1):e0089724. doi: 10.1128/spectrum.00897-24. Epub 2024 Nov 22. PMID 39576120
- [Derived] Benevolo M, Mancuso P, Allia E, Gustinucci D, Bulletti S, Cesarini E, Carozzi FM, Confortini M, Bisanzi S, Rubino T, Rollo F, Marchi N, Farruggio A, Pusiol T, Venturelli F, Giorgi Rossi P; New Technologies for Cervical Cancer 2 (NTCC2) Working Group. Determinants of p16/Ki-67 adequacy and positivity in HPV-positive women from a screening population. Cancer Cytopathol. 2021 May;129(5):383-393. doi: 10.1002/cncy.22385. Epub 2020 Nov 3. PMID 33142029